CLINICAL TRIAL: NCT04754867
Title: Pre-Test of For the Future Self: A Behavioral Intervention to Increase Success in a Smoking Cessation Program
Brief Title: Pre-Test of For the Future Self and Smoking Cessation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never initiated. PI has left the institution.
Sponsor: Carnegie Mellon University (Other)
Collaborators: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY2016_00000551
Record Dates: First submitted 2017-09-20; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Adherence, Medication
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Investigators will recruit participants planning to begin using nicotine patches in local smoking cessation programs, and randomly assign them to one of three conditions: 1) "discontinued-smoker" age-progressed future self virtual reality images vs. 2) "discontinued-smoker" + "continued smoking" age-progressed future self virtual reality images vs. 3) control - current self virtual reality images.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "discontinued-smoker" age-progressed (Experimental): Participants in the "discontinued smoker" age-progressed virtual reality condition will see two rendering of themselves in optimal health twenty years into the future, a frontal and profile view.
  Interventions: Behavioral: Future Self Virtual Reality Image - Normal Aging; Behavioral: Letter - 20 years
- "discontinued-smoker" + "continued smoking" age-progressed (Experimental): Participants in the "discontinued smoker" + "continued smoking" age-progressed virtual reality condition will see two frontal renderings of themselves twenty years in the future, one in optimal health and one incorporating appearance-related medical consequences of moderate-heavy smoking over twenty years (e.g., skin that is dry and discolored, increased wrinkles, etc.).
  Interventions: Behavioral: Future Self Virtual Reality Image - Normal Aging; Behavioral: Future Self Virtual Reality Image - Smoking Consequences Aging; Behavioral: Letter - 20 years
- Current self virtual reality images (Experimental): Participants in the current self virtual reality condition will see their present age self in a virtual reality rendering.
  Interventions: Behavioral: Current Self Virtual Reality Image; Behavioral: Letter - 3 months

INTERVENTIONS:
Behavioral: Future Self Virtual Reality Image - Normal Aging — Using software developed for this purpose, a current photograph of the subject will be aged and presented through a visual medium. The image (face) will be rendered as a 3D virtual reality avatar.
  Arms: "discontinued-smoker" + "continued smoking" age-progressed; "discontinued-smoker" age-progressed
Behavioral: Future Self Virtual Reality Image - Smoking Consequences Aging — Using software developed for this purpose, a current photograph of the participant will be aged showing the results of continued smoking and presented through a visual medium. The image (face) will be rendered as a 3D virtual reality avatar.
  Arms: "discontinued-smoker" + "continued smoking" age-progressed
Behavioral: Current Self Virtual Reality Image — Using software developed for this purpose, a current photograph of the participant will be rendered as a 3D virtual reality avatar.
  Arms: Current self virtual reality images
Behavioral: Letter - 20 years — Participants will write a 200-300 word letter to the self they see in that image in 20 years' time. The instructions will read: "Think about who you will be in 20 years from now, and write about the person you are now. What things are important and dear to you, and how do you see your life?"
  Arms: "discontinued-smoker" + "continued smoking" age-progressed; "discontinued-smoker" age-progressed
Behavioral: Letter - 3 months — Participants will write a 200-300 word letter to the self they see in that image. The instructions will read: "Think about who you will be in 3 months from now, and write about the person you are now. What things are important and dear to you, and how do you see your life?"
  Arms: Current self virtual reality images

SUMMARY:
The goal of this experimental research is to increase adherence to a smoking cessation patch among Pittsburgh residents who are trying to quit smoking. The literature on smoking cessation shows that there is a significant problem with adherence when using a transdermal patch as a nicotine replacement treatment. Less than half of patients use the patch as prescribed and adherence suffers a rapid decline during the first six weeks of treatment (Waldroup, Gifford, & Kalra, 2006). Recent work in psychology demonstrates that being more connected to our "future selves" enables better long-term decision making, in part by making future rewards more salient (and making present rewards less so). To test whether a future selves intervention might facilitate patch adherence in a smoking cessation program, investigators will recruit participants planning to begin using nicotine patches in local smoking cessation programs, and randomly assign them to one of three conditions: 1) "discontinued-smoker" age-progressed future self virtual reality images vs. 2) "discontinued-smoker" + "continued smoking" age-progressed future self virtual reality images vs. 3) control - current self virtual reality images.

DETAILED DESCRIPTION:
Several factors are thought to be relevant to the level of adherence such as the initial level of nicotine addiction (Orleans et al., 1994), gender (Gritz, Nielsen, & Brooks, 1996), concerns over weight gain due to smoking cessation (Fagerström, 2002) and side effects (Burns & Levinson, 2008). On the other hand, combining nicotine replacement treatment with behavioral therapy has been shown to improve adherence and overall abstinence (Cooper et al., 2004) and motivation is found to be an important factor related to patch use (Alterman, Gariti, Cook, & Cnaan, 1999).

Can a more vivid connection to an individual's future self facilitate smoking cessation? While behavioral interventions that enhance connection to the future self have been proven effective at mitigating present bias, they have so far been done in domains that require self-restraint (e.g., delinquency). Smoking cessation does in part require restraint, but a cessation program utilizing the nicotine patch also requires proactive daily commitment and action. Little research has been done to establish the effectiveness of a future selves intervention on behaviors that require proactive action.

Recent work in psychology demonstrates that being more connected to our "future selves" enables better long-term decision making, in part by making future rewards more salient (and making present rewards less so). To test whether a future selves intervention might facilitate patch adherence in a smoking cessation program, investigators will recruit participants planning to begin using nicotine patches in local smoking cessation programs, and randomly assign them to one of three conditions: 1) "discontinued-smoker" age-progressed future self virtual reality images vs. 2) "discontinued-smoker" + "continued smoking" age-progressed future self virtual reality images vs. 3) control - current self virtual reality images. Participants in the "discontinued smoker" age-progressed virtual reality condition will see two rendering of themselves in optimal health twenty years into the future, a frontal and profile view; participants in the "discontinued smoker" + "continued smoking" age-progressed virtual reality condition will see two frontal renderings of themselves twenty years in the future, one in optimal health and one incorporating appearance-related medical consequences of moderate-heavy smoking over twenty years (e.g., skin that is dry and discolored, increased wrinkles, etc.); participants in the current self virtual reality condition will see their present age self in a virtual reality rendering. Participants in all conditions will write a 200-300 word letter to themselves (in the treatment condition, the letter is written to their self in 20 years; in control, the letter is written to themselves in 3 months). The investigators will measure the impact of the behavioral intervention on participants' expected efficacy with smoking cessation, self-reported patch adherence, and smoking cessation success 2 and 8 weeks later.

The investigators will collect self-reported and non-invasive physiological adherence data over the course of 8 weeks on participants' adherence to the nicotine patch (self-report) and success with smoking cessation (self-report and CO analysis). For those participants self-reporting zero cigarettes smoked in the 7 day period before lab visits, investigators will administer a breath CO assessment (a simple procedure where the participant breathes into a tube and the device analyzes how many carbon dioxide parts per million are in the breath). The investigators will also asks participants if they would be willing to receive an email invitation to an online, 3-question, 6-month follow-up survey to occur four months after their last in-person visit to the laboratory.

The data collected will not be tied to identifiers; it will be used in statistical analyses assessing the effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Considering enrollment or recently enrolled (within 1 week) in one of the three designated smoking cessation programs

Exclusion Criteria:

* Use of any form of tobacco other than cigarettes
* Use of nicotine gum
* History of alcohol or drug dependency

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Adherence at two weeks | Two weeks after initial intervention
  In the past 2 weeks, how often did you wear a nicotine patch?
Adherence at eight weeks | Eight weeks after initial intervention
  In the past 2 weeks, how often did you wear a nicotine patch?

SECONDARY OUTCOMES:
Abstinence at two weeks | Two weeks after initial intervention
  In the past 2 weeks, how often did you smoke a cigarette?
Abstinence at eight weeks | Eight weeks after initial intervention
  In the past 2 weeks, how often did you smoke a cigarette?
CO ppm at two weeks | Two weeks after initial intervention
  Subjects will blow into CO analyzer.
CO ppm at eight weeks | Eight weeks after initial intervention
  Subjects will blow into CO analyzer.

IPD SHARING:
Plan to Share IPD: No